CLINICAL TRIAL: NCT02164019
Title: A Randomized Trial to Assess Patient Quality of Life and Function After Alternative Surgeries for Pathologic Fractures of
Brief Title: A Randomized Trial to Assess Patient Quality of Life and Function After Alternative Surgeries for Pathologic Fractures of the Femur
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: State University of New York - Upstate Medical University (Other); Spectrum Health Medical Group (Unknown); University of Rochester (Other); Mayo Clinic (Other); Walter Reed National Military Medical Center (U.S. Federal Agency); Duke University (Other); Montefiore Medical Center (Other); Medical University of Graz (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12-287
Record Dates: First submitted 2014-06-12; First posted 2014-06-16 (Estimated); Last update posted 2025-07-03 (Actual); Status verified 2025-07

CONDITIONS: Proximal Femoral Metastases
Keywords: Pathologic Fractures; hip replacements; 12-287
MeSH Terms: conditions — Fractures, Spontaneous | interventions — Fracture Fixation, Intramedullary; Surveys and Questionnaires

ARMS (2):
- long-stem cemented hemiarthroplasty (LSCH) (Active Comparator): (LSCH), "Hip, Ball, Rod and Cement" Replace the ball of the hip joint with a metal ball and a rod that is placed inside the thigh bone with cement to keep the implant in place. The study participation period for each patient is 360 days from the date of surgery and includes 5 defined timepoints that include the suture removal visit at 3 weeks and follow-up clinical visits for radiographs and rehabilitation progress checks at 6 weeks, 12 weeks, 6 months, and 12 months after surgery. At each follow-up visit, a combination of questionnaires and physical tests will be administered to assess physical function, general health status, disability level, and pain control. Some patients may be in a rehabilitation center or on hospice care and will miss their follow-up appointments. To collect data for the primary endpoint, the 6 week and/or 12 week TESS can be done over phone if necessary.
  Interventions: Procedure: long-stem cemented hemiarthroplasty (LSCH); Behavioral: questionnaires
- intramedullary nailing (IMN) (Active Comparator): Intramedullary nailing (IMN), "Rod and Screws" A metal rod is placed inside your thigh bone and secured in place by metal screws just below the hip and above the knee. The study participation period for each patient is 360 days from the date of surgery and includes 5 defined timepoints that include the suture removal visit at 3 weeks and follow-up clinical visits for radiographs and rehabilitation progress checks at 6 weeks, 12 weeks, 6 months, and 12 months after surgery. At each follow-up visit, a combination of questionnaires and physical tests will be administered to assess physical function, general health status, disability level, and pain control. Some patients may be in a rehabilitation center or on hospice care and will miss their follow-up appointments. To collect data for the primary endpoint, the 6 week and/or 12 week TESS can be done over phone if necessary.
  Interventions: Procedure: intramedullary nailing (IMN); Behavioral: questionnaires

INTERVENTIONS:
Procedure: long-stem cemented hemiarthroplasty (LSCH)
  Arms: long-stem cemented hemiarthroplasty (LSCH)
Procedure: intramedullary nailing (IMN)
  Arms: intramedullary nailing (IMN)
Behavioral: questionnaires

SUMMARY:
The purpose of this study is to look at two different types of surgeries regularly used for treating cancer that has spread to and weakened the thigh bone (femur). Because it is not known which of these surgeries is best, the investigators will compare the results of the two procedures. They are looking to see if differences exist (after surgery) in function, quality of life, pain control, and possible complications.

ELIGIBILITY:
Inclusion Criteria:

* Surgeon's estimated survival ≥ 1 month
* Patients presenting for orthopaedic evaluation with a painful impending pathologic femur fracture or displaced pathologic femur fracture in the intertrochanteric, pertrochanteric, or subtrochanteric region of the proximal femur. The anatomic region of interest is defined by a line drawn from the base of the femoral neck to 5 cm below the base of the lesser trochanter or 2 diaphyseal shaft widths, whichever is greater.
* Patients with an impending fracture who have had bevacizumab are eligible provided there will be a 3-week window between their last infusion and surgery.
* Diagnosis of widespread visceral and/or osseous metastatic disease based on clinical and radiographic evidence. (Patients may continue on study if surgery shows a non-malignant process.)
* All cancer diagnoses, except lymphoma, will be eligible

Exclusion Criteria:

* Estimated survival <1 month
* A large soft tissue mass or other disease involving an area outside of the defined pertrochanteric anatomic region described above. (Patients excluded based on intraoperative findings will be replaced on the study.)
* Prior surgical treatment of the area (i.e., revision cases). A biopsy does not constitute prior surgical treatment.
* Radiographic evidence of an intramedullary occlusion by blastic metastases that would necessitate an alternative method of treatment, such as a plate/screw construct.
* Diagnosis of lymphoma
* Age < 18 years
* Patients with advanced hip arthritis on radiographic imaging
* Previous randomization for a contralateral procedure as part of this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2014-06 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
differences in postoperative functional outcomes | 12 weeks
  Implant-specific differences in postoperative functional outcomes will be determined throughout the study period using Toronto Extremity Salvage Score (TESS); the primary outcome assessment will take place at the 12-week follow-up visit.

SECONDARY OUTCOMES:
postoperative complications | 1 year
  Complications will be summarized by type (e.g., superficial infection, deep infection, dislocation, etc), and complication rates will be compared between groups using Fisher's Exact test.
differences in transfusion volume | first two weeks post surgery
  The number of units of transfused blood during the first two weeks post surgery will be summarized and compared between groups using the Wilcoxon rank sum test.

CONTACTS AND LOCATIONS:
Overall Officials: John Healey, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (6):
- United States (6):
  - Spectrum Health Medical Group, Grand Rapids, Michigan
  - Memorial Sloan Kettering Cancer Center 1275 York Avenue, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - SUNY Upstate Medical University, Syracuse, New York
  - Montefiore Medical Center, The Bronx, New York
  - Duke University, Durham, North Carolina

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/